CLINICAL TRIAL: NCT06495515
Title: Efficacy and Safety of Dalpiciclib Plus Toremifene in the Treatment of Advanced First-line HR Positive and HER2 Negative Breast Cancer: a Multicenter, Single Arm, Exploratory Phase II Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tianjin Cancer Hospital...
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: CANCER; BRAEST CANCER; Late Frontline
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Trial medication/treatment:
  1. Dalpiciclib : 150mg orally, once a day, taken for 3 weeks, stopped for 1 week, with a cycle of 4 weeks. It is recommended to take medication at the same time every day, with warm water for delivery. It is recommended to do so on an empty stomach and fast for at least 1 hour before and after taking the medication.
  2. Toremifen: 60mg orally, once a day If it is a premenopausal or perimenopausal patient, it is necessary to combine with OFS (OFS includes bilateral ovariectomy or GnRHa drugs).
  The subjects will be treated according to the study protocol until disease progression, intolerable toxicity, withdrawal of informed consent, or termination of medication as determined by the researcher
  Interventions: Drug: Dalpiciclib，Toremifen

INTERVENTIONS:
Drug: Dalpiciclib，Toremifen — 1. Dalpiciclib : 150mg orally, once a day, taken for 3 weeks, stopped for 1 week, with a cycle of 4 weeks. It is recommended to take medication at the same time every day, with warm water for delivery. It is recommended to do so on an empty stomach and fast for at least 1 hour before and after taking the medication.
  2. Toremifen: 60mg orally, once a day If it is a premenopausal or perimenopausal patient, it is necessary to combine with OFS (OFS includes bilateral ovariectomy or GnRHa drugs).

SUMMARY:
Experimental population:Advanced first-line HR+, HER2 metastatic breast cancer patients

Research endpoint:

Main research endpoint:

PFS evaluated by researchers (according to RECIST 1.1 standard)

Secondary study endpoint:

ORR、CBR、DCR、OS The incidence of adverse events (AE) and severe adverse events (SAE)

Exploratory study endpoint:

Tumor infiltrating lymphocytes (sTIL) Peripheral blood lymphocyte ratio Distribution of fecal microbiota Research overall design:This study adopts a prospective, single arm design, and plans to include 36 postmenopausal or premenopausal/perimenopausal patients with metastatic breast cancer who are HR positive and HER2 negative, and receive maintenance treatment with darcy plus toremifene. In this study, the screening period did not exceed 28 days. After completing the screening examination and evaluation, eligible subjects entered the study treatment period and received maintenance treatment with darcilib combined with toremifen, for a period of 4 weeks until disease progression, intolerable toxicity, withdrawal of informed consent, or termination of medication as determined by the investigator. Conduct research according to the plan regulations Treatment and visits. Perform tumor imaging evaluation every 2 cycles (8 weeks ± 7 days) during the first 13 treatment cycles (52 weeks) of the treatment period; Afterwards, tumor imaging evaluation will be conducted every 3 cycles (12 weeks ± 7 days). Subjects should visit the research center at the end of treatment/withdrawal from the study to complete corresponding safety checks and imaging evaluations; And visit the research center 28 days after the last treatment to complete the corresponding safety assessment.

DETAILED DESCRIPTION:
Inclusion Criteria :

Participants must meet all of the following inclusion criteria in order to be enrolled in this trial:

1. Postmenopausal or premenopausal/perimenopausal female patients aged ≥ 18 years and ≤ 75 years old,

   Meet one of the following conditions:

   a) Previously underwent bilateral oophorectomy, or aged ≥ 60 years old; or b) Age<60, natural postmenopausal state (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without any other pathological or physiological reasons), E2 and FSH at postmenopausal levels.

   c) Premenopausal or perimenopausal female patients can also be selected, but they must be willing to receive LHRH agonist treatment during the study period.
2. ECOG PS 0-1；
3. Female breast cancer patients diagnosed as HR positive and HER2 negative by pathology have evidence of local recurrence or metastasis, which is not suitable for surgical resection or radiotherapy for the purpose of cure.

It has been diagnosed as HR positive and HER2 negative breast cancer (ER and PR ≥ 10%)

HER2 is negative. If HER2 is expressed as 2+, in situ hybridization testing is required to confirm that the HER2 gene has not been amplified; 4. The patient's previous endocrine therapy must meet the following conditions:

A) Late stage: did not receive any endocrine therapy; Progression within 12 months of receiving other endocrine treatments (except tamoxifen) in the late stage; b) Stage of adjuvant endocrine therapy: Progress over 12 months after completion of tamoxifen assisted endocrine therapy; During the use of aromatase inhibitors (treatment duration exceeding 6 months) or after completion of treatment, progress may occur.

According to the RECIST 1.1 standard, there should be at least one measurable lesion present or only bone metastases (including osteolytic lesions or mixed osteolytic/osteogenic lesions).

6. The functional level of organs must meet the following requirements:

1. Blood routine

   •ANC≥1.5×109/L；

   •PLT≥90×109/L；

   •Hb≥90 g/L；
2. Blood biochemistry

   * TBIL≤1.5×ULN； ALT and AST ≤ 2 × ULN;
   * BUN and Cr ≤ 1.5 × ULN with creatinine clearance rate ≥ 50 mL/min (Cockcroft Gault formula);
3. Cardiac color Doppler ultrasound

   •LVEF≥50%；
4. 12 lead electrocardiogram The QT interval (QTcF) corrected by the Fridericia method is<470 ms for females.

7. Patients with negative serum pregnancy test and potential fertility must agree to use it during treatment and on the last attempt Use effective non hormonal contraceptive methods for at least 12 months after the trial drug.

8. Voluntarily participate in this study, sign informed consent, have good compliance, and are willing to cooperate with follow-up.

Exclusion criteria:

1. The previous pathological diagnosis was HER2 positive breast cancer.
2. Researchers determine patients who are not suitable for endocrine therapy. This includes late stage patients who have symptoms, have spread to the internal organs, and are at risk of life-threatening complications in the short term (including patients with uncontrollable exudates (chest, pericardium, abdominal cavity) through drainage or other methods, pulmonary lymphangitis, and more than 50% liver involvement).
3. The patient has undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or has not fully recovered from such surgical procedures.
4. Patients with extensive advanced/metastatic, symptomatic visceral diseases, or known uncontrolled or symptomatic brain metastases.
5. Previously used any CDK inhibitors, tamoxifen, everolimus, or drugs that inhibit the PI3K mTOR pathway for treatment. Using strong or moderate CYP3A4 and/or CYP2D6 inhibitors or inducers.
6. Other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
7. Have suffered from any heart disease, including: (1) angina pectoris; (2) Arrhythmias that require medication treatment or have clinical significance; (3) Myocardial infarction; (4) Heart failure; (5) Any other heart disease determined by the researcher as unsuitable for participation in this trial.
8. Inability to swallow, intestinal obstruction, or other factors that affect medication administration and absorption.
9. Known to be allergic to darcilib, letrozole, or any excipients.
10. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial period.
11. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
12. There are other serious physical or mental illnesses or laboratory test abnormalities that may increase the risk of participating in the study, interfere with the research results, and any other circumstances that the researcher deems unsuitable for participation in this study.

Termination of treatment criteria:

1. Discovering unexpected, significant, or unacceptable risks to the subjects;
2. During the execution of the experiment, significant errors were found in the plan;
3. The research drug/trial treatment is ineffective, or continuing the trial is meaningless;
4. Due to factors such as severe delay in subject selection or frequent protocol deviations, it is extremely difficult to complete the experiment;
5. The subjects experienced severe adverse events, which were intolerable and could not be relieved;
6. The subject decides to withdraw on their own;
7. The subjects have poor compliance with the research protocol;

Trial medication/treatment:

1. Dalpiciclib : 150mg orally, once a day, taken for 3 weeks, stopped for 1 week, with a cycle of 4 weeks. It is recommended to take medication at the same time every day, with warm water for delivery. It is recommended to do so on an empty stomach and fast for at least 1 hour before and after taking the medication.
2. Toremifen: 60mg orally, once a day If it is a premenopausal or perimenopausal patient, it is necessary to combine with OFS (OFS includes bilateral ovariectomy or GnRHa drugs).

The subjects will be treated according to the study protocol until disease progression, intolerable toxicity, withdrawal of informed consent, or termination of medication as determined by the researcher 8. Disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal or premenopausal/perimenopausal female patients aged ≥ 18 years and ≤ 75 years old,

   Meet one of the following conditions:

   a) Previously underwent bilateral oophorectomy, or aged ≥ 60 years old; or b) Age<60, natural postmenopausal state (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without any other pathological or physiological reasons), E2 and FSH at postmenopausal levels.

   c) Premenopausal or perimenopausal female patients can also be selected, but they must be willing to receive LHRH agonist treatment during the study period.
2. ECOG PS 0-1；
3. Female breast cancer patients diagnosed as HR positive and HER2 negative by pathology have evidence of local recurrence or metastasis, which is not suitable for surgical resection or radiotherapy for the purpose of cure.

It has been diagnosed as HR positive and HER2 negative breast cancer (ER and PR ≥ 10%)

HER2 is negative. If HER2 is expressed as 2+, in situ hybridization testing is required to confirm that the HER2 gene has not been amplified; 4. The patient's previous endocrine therapy must meet the following conditions:

A) Late stage: did not receive any endocrine therapy; Progression within 12 months of receiving other endocrine treatments (except tamoxifen) in the late stage; b) Stage of adjuvant endocrine therapy: Progress over 12 months after completion of tamoxifen assisted endocrine therapy; During the use of aromatase inhibitors (treatment duration exceeding 6 months) or after completion of treatment, progress may occur.

According to the RECIST 1.1 standard, there should be at least one measurable lesion present or only bone metastases (including osteolytic lesions or mixed osteolytic/osteogenic lesions).

6. The functional level of organs must meet the following requirements:

1. Blood routine

   •ANC≥1.5×109/L；

   •PLT≥90×109/L；

   •Hb≥90 g/L；
2. Blood biochemistry

   * TBIL≤1.5×ULN； ALT and AST ≤ 2 × ULN;
   * BUN and Cr ≤ 1.5 × ULN with creatinine clearance rate ≥ 50 mL/min (Cockcroft Gault formula);
3. Cardiac color Doppler ultrasound

   •LVEF≥50%；
4. 12 lead electrocardiogram The QT interval (QTcF) corrected by the Fridericia method is<470 ms for females.

7. Patients with negative serum pregnancy test and potential fertility must agree to use it during treatment and on the last attempt Use effective non hormonal contraceptive methods for at least 12 months after the trial drug.

8. Voluntarily participate in this study, sign informed consent, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. The previous pathological diagnosis was HER2 positive breast cancer.
2. Researchers determine patients who are not suitable for endocrine therapy. This includes late stage patients who have symptoms, have spread to the internal organs, and are at risk of life-threatening complications in the short term (including patients with uncontrollable exudates (chest, pericardium, abdominal cavity) through drainage or other methods, pulmonary lymphangitis, and more than 50% liver involvement).
3. The patient has undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or has not fully recovered from such surgical procedures.
4. Patients with extensive advanced/metastatic, symptomatic visceral diseases, or known uncontrolled or symptomatic brain metastases.
5. Previously used any CDK inhibitors, tamoxifen, everolimus, or drugs that inhibit the PI3K mTOR pathway for treatment. Using strong or moderate CYP3A4 and/or CYP2D6 inhibitors or inducers.
6. Other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
7. Have suffered from any heart disease, including: (1) angina pectoris; (2) Arrhythmias that require medication treatment or have clinical significance; (3) Myocardial infarction; (4) Heart failure; (5) Any other heart disease determined by the researcher as unsuitable for participation in this trial.
8. Inability to swallow, intestinal obstruction, or other factors that affect medication administration and absorption.
9. Known to be allergic to darcilib, letrozole, or any excipients.
10. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or those in the whole family Female patients of childbearing age who were unwilling to take effective contraceptive measures during the trial period.
11. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
12. Other serious physical or mental illnesses or laboratory test abnormalities may increase the risk of participating in the study, or Disturb the research results and any other circumstances that the researcher deems unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 30.6 months
  The time from randomization to disease progression evaluated by researchers for patients

IPD SHARING:
Plan to Share IPD: No